CLINICAL TRIAL: NCT04553575
Title: Follow-up CoViD-19 Patients Hospitalized in Reims University Hospital Between the 01/03/2020 and 30/04/2020
Brief Title: CoViD-19 Patient in Reims University Hospital in March to April 2020
Acronym: COVID-Reims
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PO20124*
Record Dates: First submitted 2020-09-15; First posted 2020-09-17 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Coronavirus Infections
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CoViD-19 patients cohort: Patients are followed for 2 years after diagnosis. The only one intervention is blood samples withdrawn for serologies
  Interventions: Biological: serology

INTERVENTIONS:
Biological: serology — biological blood samples withdrawn at 6, 12 and 24 months

SUMMARY:
Medical context: Follow-up of a retrospective cohort of 499 cases of CoViD-19, hospitalized at the University Hospital of Reims during the health crisis, prospectively up to two years of follow-up.

Possible intervention for serological monitoring, leading to a change from category 3 to category 2 (French law on human person research)

Aim of the study: To know the factors of gravity of CoViD-19, to know its prognostic factors, to see how the evolution of the treatments implemented have influenced the fate of the patients.

Material and methods:

Type of study: cohort study Population: Patients in the CoViD-19 cohort - Reims Calendar: September 2020 - July 2022

Expected results: Better knowledge of the cares of patients with CoViD-19

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalized for CoViD-19 infection during the health crisis, in a short-stay service of Reims University Hospital and included in Covid-19 Cohort
* Age > 18 years
* Patient who benefit from the national health insurance coverage
* patient agree for participation (consent form signed)

Exclusion Criteria:

* Patient protected by law

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient hospitalized for CoViD-19 infection during the health crisis, in a short-stay service of Reims University Hospital and included in Covid-19 Cohort
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2022-05-24 (Actual); Study Completion 2022-08-04 (Actual)

PRIMARY OUTCOMES:
Health status in the 2 years after CoViD-19 diagnosis | 2 years follow up
  status : dead or alive persistante respiratory distress (yes / no)

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France